CLINICAL TRIAL: NCT02650583
Title: Enhancing Connections Program in Palliative Care: Taking Care of the Children
Brief Title: Enhancing Connections Program in Improving Communication Between Patients With Incurable Cancer and Their Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 9480; NCI-2015-01941 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9480 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2015-12-11; First posted 2016-01-08 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Advanced Malignant Neoplasm
MeSH Terms: interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Supportive care (Enhancing Connections Program) (Experimental): Patients participate in Enhancing Connections Program comprising of anchoring patients to help their child, adding to listening skills, building on listening skills, being a detective of their child's coping, and celebrating success for 5 sessions. Patients also receive workbook which includes text from the sessions, handouts, and at-home assignments to be completed between sessions.
  Interventions: Other: Educational Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Receive Enhancing Connections Program
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies the use of the Enhancing Connections Program in improving communication between patients with incurable cancer and their children. The Enhancing Connections Program is an educational program that may provide patients with new competencies to improve communication with their children and help them to cope with their parent's incurable cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the feasibility of the study protocol in advanced cancer patients (recruitment/retention, dosage and fidelity of the intervention; program acceptability of program; and logistics).

II. To evaluate the short-term impact of the program on the diagnosed parents' and children's adjustment using a within group design (pre- and post-test design).

III. To compare outcomes from the Enhancing Connections Program with outcomes obtained from the completed Phase III trial (between group design).

OUTLINE:

Patients participate in Enhancing Connections Program comprising of anchoring patients to help their child, adding to listening skills, building on listening skills, being a detective of their child's coping, and celebrating success for 5 sessions. Patients also receive workbook which includes text from the sessions, handouts, and at-home assignments to be completed between sessions.

ELIGIBILITY:
Inclusion Criteria:

* Parents will be eligible if they have a diagnosis of incurable cancer of any type
* Read and write English among their languages of choice
* Have a child 5-17 years old living at home who has been told their parent's cancer diagnosis
* The child does not have learning challenges

Exclusion Criteria:

* Parents will be excluded if they are enrolled in hospice at time of enrollment; (however, they will be allowed to continue in the study if they enroll in hospice after beginning the study)
* Parents will be ineligible if their child lives in the home less than 50% of the time

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-12-28 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Change in EC-palliative care (PC) parents' and children's scores (parent-reported) on standardized questionnaires from baseline to post-intervention | Baseline to up to 3 months
  Baseline scores will be compared with post-intervention scores on the same measures. Analysis of covariance will be used to test for significant differences between pre- and post-test scores.
Differences between the telephone-delivered and the in-person delivered program | Up to 3 months
  Linear mixed modeling based on maximum likelihood estimation will be used to test the differences between the telephone-delivered and the in-person delivered program.
Dosage and fidelity | Up to 3 months
  Will be monitored for each intervention session using the performance checklists, the same checklists used to monitor dosage and fidelity in the Enhancing Connections (EC) trial. (Each session of the Program has its own unique Performance Checklist and each item is scored from 0-2. Performance Checklist items are specific to each session of the Program to be delivered by the patient educator. Higher scores denote higher performance by the patient educator and greater confidence that the Program was delivered as designed. The Performance Checklist is only used to monitor the performance of the
Duration of intervention sessions | Up to 3 months
Number of patients recruited and retained, tracked on recruitment spreadsheets | Up to 3 months
  Three methods of recruitment will be monitored: self-referral, provider referral, and recruitment letter.
Parent and child adjustment at completion of the EC-PC program, as measured by standardized questionnaire | Up to 3 months
  Will be compared with outcomes obtained from the intervention group in the EC-RCT (historical comparison group).
Percentage of participants who complete both baseline and post-intervention sets of questionnaires with no missing data | Up to 3 months
  Assessed at baseline and post-intervention (up to 3 months).
Percentage of participants who return both baseline and post-intervention sets of questionnaires within 2 weeks of receipt | Up to 14 weeks
  Assessed at baseline and post-intervention (up to 3 months).
Program acceptability (per session, overall, duration of program, interval between intervention sessions) | At Session 5, occurring within up to 3 months
  Will be assessed from a debriefing interview in Session 5 that includes the parents' attributed gains of the program and their responses to the program's content, format, in-session, and at-home assignments.
Rate of receipt of mailed materials both to participants and from participants (e.g., signed consents, baseline data; parent's materials) | Baseline
Rate of success in scheduling and completing intervention sessions | At Session 5, occurring within up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Frances Lewis, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States